CLINICAL TRIAL: NCT05476016
Title: A Single-Centre, Open-label Study Testing the Safety and Performance of the Glyconics-SX System in Individuals With or Without Type 2 Diabetes
Brief Title: Safety and Performance of the Glyconics-SX System (ANODE02)
Acronym: ANODE02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glyconics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NIRDM-SXCIP02
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: Screening among individuals with or without known diabetes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label, single arm with identical intervention for all participants (Experimental): Glycated keratin assessed by near-infrared and glycated haemoglobin (HbA1c) assessed based on finger prick blood drop sample
  Interventions: Device: Near-infrared (NIR)

INTERVENTIONS:
Device: Near-infrared (NIR) — NIR spectral assessment of glycated nail keratin vs HbA1c
  Other Names: point-of-care device (HbA1c analyser)

SUMMARY:
The main clinical study objective is to retrieve initial high quality spectra measurements indicative of the accuracy of the Glyconics-SX System in distinguishing between individuals with or without T2DM based on known and/or assumed clinical status and as controlled by values of an internal biomarker indicative of glycaemia, HbA1c, as measured with a validated comparator device.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adults (≥18 years of age) with known or unknown T2DM status willing to participate in and provide a written consent for the study
* willingness to undertake assisted assessment of glycaemia by both the NIR spectra measurement, and HbA1c by finger prick test
* Individuals with two visually assessed apparently healthy, undamaged, and intact fingernails, one in both right- and left-hand middle fingers

Exclusion Criteria:

Individuals with any known medical conditions impacting either of the assessment methodology for glycaemia, such as

* anaemia (iron deficiency sickle cell anaemia or similar)
* haemoglobinopathies or atypical haemoglobin subtypes not detectable by regular assays,
* severe renal impairment (CKD stage III-IV) or decompensated hepatic disease
* severe Vitamin D deficiency
* known severe immunodeficiency such as HIV, malignancy or other chronic condition significantly impacting assessment of glycaemia
* eating disorders (as per clinical assessment)
* Recent (within 28 days) blood donation

  o Any structural, deviating and visually detectable deviations in the appearance of the nails potentially impacting the spectra measurement, including
* nail dystrophy or deformity
* severe nail infections (onychomycosis causing visual changes in the appearance of the nail)
* rare hereditable conditions impacting the structure of keratin
* mechanical damage or marks on the surface of the nail after removal of nail polish
* use of acrylic or gel nail decoration and polish, which cannot be removed o Any systemic or topical medication known to modify either the surface or structure of the nail or accuracy of HbA1c value.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Glyconics-SX System in detection of DM status based on dichotomised outcomes as per the chemometric model (HbA1c measurements as internal control) | 60 seconds
  Overall probability of correct classification by the chemometric model output (yes / no DM)

SECONDARY OUTCOMES:
Assessment of sensitivity and specificity for chemometric model outcomes | 60 seconds
  False positive and false negative assessments in %
Calculation of negative and positive predictive value for the chemometric model | 60 seconds
  Calculated values in %
Calculation of AUC with axis defined by false positive and negative rates for the model | 60 seconds
  Area under curve
Median (IQR) HbA1c values in both groups (with or without DM) | 4 minutes
  HbA1c value in mmol/mol
Analysis of safety outcomes, included suspected de novo DM diagnosis based on HbA1c | 15 minutes
  adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Sant Marti, Barcelona, Spain